CLINICAL TRIAL: NCT00720928
Title: A Multi-Center, Prospective Single Arm Study to Assess the Efficacy and Safety of RETISERT (Intravitreal Flucinolone Acetonide 0.59mg) in Patients With Refractory Ocular Behcet's Disease
Brief Title: Flucinolone Acetonide Implant for Treating Refractory Ocular Behcet's Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Seoul National University Hospital (Other); Kyunghee University Medical Center (Other)
Responsible Party: Young Hee Yoon, MD/Professor and Chairman, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-2008-1
Record Dates: First submitted 2008-07-18; First posted 2008-07-23 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: Ocular Behcet's Disease,; Non-Infectious Uveitis; Refractory Uveitis
Keywords: Behcet's disease; posterior uveitis; flucinolone acetonide; RETISERT
MeSH Terms: conditions — Uveitis; Behcet Syndrome; Uveitis, Posterior | interventions — Fluocinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single group (Other): Posterior uveitis patients having complete or incomplete type of Behcet's disease; typical ocular lesion and at least, one of the main symptoms or two of the additional symptoms.
  Selection of study eye : For patients with unilateral uveitis, the study eye will be the affected eye; for patients with bilateral uveitis, the study eye will be the more severely affected eye (i.e., the eye having suffered more recurrences in the previous year, or if equal, the eye having received more therapy in the previous year, or if equal, the eye having the worse VA, or if equal, the eye clinically judged to be the more severely affected eye).
  Interventions: Drug: flucinolone acetonide

INTERVENTIONS:
Drug: flucinolone acetonide — Intra-vitreal implantation of RETISERT on the study eye. The implant is a sustained-release delivery system containing 0.59 mg of flucinolone acetonide designed to deliver the drug for approximately 3 years.
  Other Names: RETISERT

SUMMARY:
Objectives:

To describe the safety and efficacy of intravitreal flucinolone acetonide implants in the management of patients having refractory ocular Behcet's disease

Hypothesis:

A descriptive observational study

Study design:

A 1-year, multi-center (including four Korean medical centers) observational study

DETAILED DESCRIPTION:
A multi-center, prospective single arm study to assess the efficacy and safety of retisert (intravitreal flucinolone acetonide 0.59 mg) in patients with refractory ocular Behcet's disease. This study will be conducted at 4 sites, located in Korea. The number of subject is expected approximately 15 patients. The medical records for the patients meeting following inclusion/exclusion criteria will be collected until 1 year after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females at least 18 years of age having complete or incomplete type of Behcet's disease according to the revised diagnostic criteria proposed by the Behcet's Disease Research Committee of Japan in 2003; typical ocular lesion and at least, one of the main symptoms or two of the additional symptoms.
* One or both eyes having a history of recurrent or chronic ocular Behcet's disease affecting the eye more than 1 year duration requiring either systemic corticosteroid or other equivalent systemic therapy for at least three months prior to enrollment; OR at least 2 sub-Tenon's injections of corticosteroid for the management of uveitis during the six months prior to enrollment; OR at least 2 separate recurrences within the six months prior to enrollment requiring either systemic corticosteroid therapy or sub-Tenon's injection of corticosteroids
* At the time of enrollment the implanted eye must have: ≤ 10 anterior chamber cells/HPF and a vitreous haze ≤ grade 2
* Visual acuity of at least 1.4 logMAR units (Snellen 20/500).

Exclusion Criteria:

* Allergy to FA or any component of the delivery system
* History of only posterior segment uveitis not accompanied by vitritis or macular edema
* History of iritis only and no vitreous cells or vitreous haze
* Uveitis with infectious etiology
* Vitreous hemorrhage
* Presence of a toxoplasmosis scar in the study eye
* Peripheral retinal detachment in area of implantation
* Media opacity precluding evaluation of the retina and vitreous
* Uncontrolled increased intraocular pressure(IOP)(>21mmHg)at the time of retisert implantation
* Ocular surgery on the study eye within 3 months prior to enrollment
* Patients requiring chronic systemic corticosteroid therapy (>15mg prednisone daily) or systemic immunosuppressive therapy to manage non-ocular disease
* Patients who have tested positive for human immunodeficiency virus
* Pregnant or lactating females
* Females of childbearing potential considering becoming pregnant during the course of the study and those not taking effective contraception/precautions to avoid pregnancy
* Patients for whom, in the physician's opinion, any of the protocol procedures may pose a special risk not outweighed by the potential benefits of participating in the study
* Patients who are unlikely to comply with the study protocol or who are likely to be moving and lost to follow-up in the 1 year
* Patients who are currently enrolled in any other IND or investigational study or who have participated in an IND or investigational study within 1 month of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-12 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Recurrence in the 36 wks, with one or more of the following events ->2 step Increase in the number of cells in the A/C -2 step increase in the vitreous haze -deterioration in visual acuity | 1 year

SECONDARY OUTCOMES:
Post-implantation recurrence of uveitis rate: within-patient comparison of responding eyes (implant vs. fellow)and etc. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Young Hee Yoon, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea